CLINICAL TRIAL: NCT03637036
Title: An Improvement Project to Evaluate the Effectiveness of Different Reminders Designed to Increase the University Hospitals Birmingham NHS Foundation Trust's Staff Uptake of the Seasonal Influenza Vaccine
Brief Title: An Improvement Project Around Staffs' Influenza Vaccine Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warwick (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Principal Investigator, Professor Richard Lilford, Professor of Public Health, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RRK6479
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants receive one of four types of communications inviting them to take up the influenza vaccination in a randomized fashion. Participants will not be explicitly told that alternative versions of the communications are being sent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Condition (Other): A general communication intervention will occur inviting staff to take up the influenza vaccination, without a specific authority or social norm designated.
  Interventions: Other: Communication intervention
- Authority Condition (Other): A communication intervention will occur inviting staff to take up the influenza vaccination with a specific authority but not a social norm designated.
  Interventions: Other: Communication intervention
- Norms Condition (Other): A communication intervention will occur inviting staff to take up the influenza vaccination with a social norm but not a specific authority designated.
  Interventions: Other: Communication intervention
- Authority + Norms Condition (Other): A communication intervention will occur inviting staff to take up the influenza vaccination with a specific authority and a social norm designated.
  Interventions: Other: Communication intervention

INTERVENTIONS:
Other: Communication intervention — The intervention is a communication inviting staff to take up the influenza vaccination. Different versions of the communication are created, and the investigators will compare uptake rates between staff that received different letters.

SUMMARY:
To reach seasonal vaccination against influenza targets, University Hospitals Birmingham (UHB) already invites staff to take up the vaccination, and every November reminds staff that have not yet vaccinated to do so. The current protocol describes a randomized controlled trial (RCT) in which staff will be sent different reminders, and the investigators will compare the proportion of staff that go on to vaccinate after receiving each reminder.

DETAILED DESCRIPTION:
Seasonal vaccination against influenza is recommended for NHS staff. , To increase vaccination rates, NHS England put forth a Commissioning for Quality and Innovation goal for the 2018/2019 season of 75%. University Hospitals Birmingham NHS Foundation Trust (UHB) wants its vaccination rate to surpass this target. Since staff get infected outside of the hospital and from patients staff vaccination does not provide significant 'herd immunity'

To reach past targets, every September UHB already invites staff to take up the vaccination, and regularly reminds staff that have not yet vaccinated to do so. The current protocol describes a randomized controlled trial (RCT) in which staff will be sent a different letter when first invited to receive vaccination, and we will compare the proportion of staff that go on to vaccinate after receiving each type of letter..

To conduct the RCT the research team will design four letter styles. One factor will emphasize an authority figure inviting staff to vaccinate (the Chief Executive, who is also a doctor). The other factor will emphasize a competitive social norm describing vaccination rates in peer hospitals, including Addenbrooke's, Cambridge University Hospitals (which has exemplary rates) see appendix A and across American hospitals (which also have high rates). Letters will be sent to staff in the first week in October by UHB's communications team and they will be disseminated in a randomized fashion.

The UoW's role in this study is to advise the study's design and write-up the project for publication. UHB will approve the reminders, send the reminders, retrieve the data, and analyse the data. No individual-level data will be transferred across organizations. All individual-level data will be managed by authorized UHB employees, e.g., a UHB statistician will randomize staff to receive different reminders and analyze the data, and UHB's communication team to disseminate the reminders.

ELIGIBILITY:
Inclusion Criteria:

* All UHB staff eligible for the seasonal influenza vaccination are eligible for this study. (no patients are included)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8438 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Vaccination uptake | 3 months
  Whether participants vaccinated (Yes, No)

SECONDARY OUTCOMES:
Vaccination uptake date | 3 months
  The date participants received vaccination (DD-MM-YYYY or blank if not vaccinated)
Vaccination uptake reflusal | 3 months
  Whether participants formally indicated refusal to vaccinate (Yes, No)
Vaccination uptake alternative location | 3
  Whether participants formally indicated being vaccinated at another location (Yes, No)

OTHER OUTCOMES:
Group number | 3 months
  This data describes what communication participants received
Worksite | 3 months
  This data describes what location within the organization participants work
Job Role | 3 months
  This data describes participants' job roles
Gender | 3 months
  This data describes participants' gender

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Lilford, Principal Investigator — University of Warwick
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust (UHB), Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03637036/Prot_SAP_001.pdf